CLINICAL TRIAL: NCT01246635
Title: A Prospective, Multi-Center, Randomized, Single-Blind, Controlled Study Comparing the Trufit CB (Cartilage Bone) Implant to Microfracture for the Treatment of Patients With Single, Isolated Defects of the Knee
Brief Title: Smith & Nephew's European Trufit Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to slow and insufficient total enrollment.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CSA-2005-02
Record Dates: First submitted 2010-11-14; First posted 2010-11-23 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Defect of Articular Cartilage
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TRUFIT CB with accelerated rehab. (Experimental)
  Interventions: Device: Trufit CB (Cartilage Bone) Implant
- TRUFIT CB with standard rehab. (Experimental)
  Interventions: Device: Trufit CB (Cartilage Bone) Implant
- • Microfracture with rehabilitation (Active Comparator)
  Interventions: Procedure: Microfracture if the knee

INTERVENTIONS:
Device: Trufit CB (Cartilage Bone) Implant — Implantation of 5,7, 9, or 11 mm Trufit CB Implants for small cartilage lesions. A maximum of two Trufit CB plugs may be implanted.
  Arms: TRUFIT CB with accelerated rehab.; TRUFIT CB with standard rehab.
Procedure: Microfracture if the knee — Creation of small holes through subchondral bone with the goal of stimulating cartilage growth
  Arms: • Microfracture with rehabilitation

SUMMARY:
The purpose of this clinical study is to demonstrate the effectiveness and safety of the Trufit CB (Cartilage Bone) implant for the treatment of single, isolated cartilage defects of the knee compared to Microfracture.

DETAILED DESCRIPTION:
Up to 315 subjects, ages 18 years and older with a single, isolated cartilage defect of the knee will be randomized in a 1:1:1 ratio to 1 of 3 treatment groups:

* Trufit CB Implant with rehabilitation protocol;
* Trufit CB Implant with rehabilitation protocol;
* Microfracture with rehabilitation protocol

Rehabilitation program may be standard (6 weeks touch weight to full weight bearing) or accelerated (2 weeks touch weight to full weight bearing).

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent;
* Eighteen (18) years or older and skeletally mature on the date of study enrollment;
* Willing and able to attend all follow up visits and complete all study related procedures and evaluations including, but not limited to adhering to the rehabilitation protocol;
* Single, isolated cartilage defect (ICRS Grade III - IV) in the knee (medial or lateral femoral condyle or trochlea) that is ≥ 1cm2 (10 mm) and ≤ 2cm2 (20 mm) in area and requiring a maximum of 2 implants (if randomized to TRUFIT CB); Note: Lesion size should be assessed as the product of the longest diameter and its perpendicular applied at the widest portion of the lesion.
* Candidate for cartilage repair surgery as a result of a single, isolated symptomatic cartilage lesion;
* Presents with stable health at the time of study enrollment;
* BMI of ≤ 32.

Exclusion Criteria:

* Female of child-bearing potential who is pregnant or plans to become pregnant over the course of the study;
* History of alcohol or drug abuse;
* Presents with patellofemoral instability or other anatomical malalignment in the study knee;
* Any diagnosis that would preclude the patient from successfully completing the study rehabilitation protocols;
* Unable or unwilling to follow post operative procedures (e.g. rehabilitation protocol);
* Received one or more intra-articular steroid injections in the study knee within the previous 3 months;
* Presents with ipsilateral hip disease, as determined by pain or restricted range of motion upon physical examination;
* Treated with either an investigational device or drug within one (1) month of study enrollment, or plans to be treated with an investigational device or drug in the next 24 months;
* Diagnosed rheumatoid arthritis, ankylosing spondylitis (Bechterew syndrome), or calcium pyrophosphate dihydrate disease(chondrocalcinosis);
* History of severe vascular or neurological disease, uncontrolled diabetes, or is immunosuppressed (e.g. HIV positive);
* Musculoskeletal disease, including degenerative bone diseases such as osteochondritis dissecans and osteonecrosis;
* Pathologic conditions of the bone (e.g. osteoporosis, cystic changes, hyperparathyroidism, Paget's Disease, hypercalcemia, prolonged use of steroids);
* Active infection, or evidence thereof, at the lesion site;
* Requires the use of any medication(s) or treatment(s) known to have an effect on bone metabolism (e.g. bisphosphonates, chemotherapeutic or immunosuppressive agents);
* Requires concomitant osteotomy, partial lateral meniscectomy or complete meniscectomy; Note: Concomitant ACL reconstruction or revision, as well as meniscal repair and partial medial meniscectomies are permitted under the study protocol.
* Has undergone an ACL reconstruction, osteotomy, chondral resurfacing procedure or partial meniscectomy (≤ central third of the meniscus) in the last year and has not completed at least 6 months of rehabilitation since such surgery; Note: Patients who have undergone these procedures within the last year and have completed at least 6 months of rehabilitation are eligible to participate in the study.
* Any active, implanted medical device (e.g. cochlear implant) or metallic implant (other then dental work) that may interfere with Magnetic Resonance Imaging (MRI);
* Any condition (e.g. claustrophobia) that may interfere with the patient's ability to undergo MRI;
* Diagnosis requiring placement of an active implant (e.g. cardiac pacemaker, vagus nerve stimulator, etc.) within the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent change in the Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline | 6 months post-procedure

SECONDARY OUTCOMES:
Percent improvement from baseline in the KOOS Knee Survey Score at all time-points | 2 weeks, 6, weeks, 3 months, (6 months - primary measure), 12 months and 24 months post-procedure
Positive change in activity level from baseline to each visit, as measured by the Tegner Activity Scale at all time-points. | 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months post-procedure
Difference in Pain Scores on the Visual Analog Scale from baseline at all post operative time-points. | 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months post-procedure
Magnetic resonance evaluation of cartilage and underlying bone using the MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) scale | 12 and 24 months post-procedure
Proportion of subjects (compared to baseline) with cartilage classifications within the four groups defined by the International Cartilage Repair Society (ICRS) scoring system | 24 months post-procedure
  Evaluation of cartilage at 24 months post-procedure will only occur for subjects who consent to a second-look biopsy.
Histological evaluation of cartilage | 24 months post-procedure
  Histological characterization of cartilage will only occur for those subjects consenting to both the second look arthroscopy and biopsy at 24-months post-procedure.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months post-procedure

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (4):
  - Karl Brabants, MD, Antwerp
  - Prof. Dr. K.F. Almqvist, Ghent
  - Toon Claes, MD, Herentals
  - Johan Vanlauwe, Leuven
- Aalborg Private Hospital A/S, Aalborg, Denmark
- Johannes Holz, MD, Hamburg, Germany
- Kevin J. Mulhall, Dublin, Ireland
- Netherlands (2):
  - Sander Koeter, MD, Nijmegen
  - Kees van Egmond, MD, Zwolle
- Lars Engebretsen, MD, Oslo, Norway
- Magnus Forssblad, MD, Stockholm, Sweden
- United Kingdom (3):
  - Angus Robertson, MD, Cardiff
  - Tim Spalding, MD, Coventry
  - David Chesney, Fife Keith